CLINICAL TRIAL: NCT02887755
Title: Assessing the Feasibility of a Novel Non-Invasive Sensor for Guiding Wounded Warrior Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 412936
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Rehabilitation Post-amputation
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amputee Group (Experimental): In this study n=20 returning US military combatants between 18 and 45 years of age who have unilateral transtibial or transfemoral amputation will be asked to perform two aerobic exercise tests while we4aring the NIRS sensor. Subjects must be medically cleared and able to complete approximately 30 minutes of physical activity.
  Interventions: Device: Near-Infrared Spectroscopy (NIRS) Sensor

INTERVENTIONS:
Device: Near-Infrared Spectroscopy (NIRS) Sensor — These sensors utilize NIRS to evaluate oxygenated and deoxygenated hemoglobin, total oxygenation index and total blood flow. This is done by bouncing infrared light off of chromatophores (located within red blood cells), which is then refracted off of the cells in the capillary beds to the topical sensor.

SUMMARY:
The purpose of this study is to test a low cost, non-invasive, wearable near-infrared spectroscopy (NIRS) sensor, previously validated for able-bodied athletes as a rehabilitation aid for war-fighters with lower extremity limb loss. This sensor can record real-time physiologic data that relates to total fitness capacity and exertion levels and may help develop individualized programs on a per-patient basis. The uniqueness of this NIRS measurement system is that it provides real-time muscular oxygenation, dehydration, and iron status during whole-body exercise, as well as training-induced adaptations. Currently, no technology like this has been tested in an amputee population. Successfully validating this technology in a wounded warrior population would provide vital information regarding tissue perfusion after injury and new opportunities for improving rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Military health care beneficiary and veterans for enrollment.
2. Between 18 and 45 year old.
3. Possess a unilateral transtibial or transfemoral amputation.
4. Low risk for cardiovascular disease.
5. Ambulatory without assistive ambulatory device.

Exclusion Criteria:

1. Exclusion criteria includes individuals outside of our age range or if over the age of 18 and under the age of 45 will be excluded if found at risk according to the ACSM/AHA pre-participation screening questionnaire for exercise testing.
2. Told by a doctor that they should not exercise.
3. Orthopedic injury/surgery of the lower extremity within the last year
4. Less than 5" x 2.5" of soft tissue proximal to the prostheses (since the sensor will need to be placed on the soft tissue proximally)
5. Hip or shoulder disarticulation.
6. Regular use of medications designed to alter cardiovascular function;
7. Unwilling to comply with the study protocol.
8. Individuals with a fat layer greater than 10mm in correspondence of the location of the NIRS probe (thigh).
9. Allergic reaction to latex, cotton, or polyester, which are the primary materials of an ace bandage.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Single Stage Treadmill Test | Single Study Visit (Study consists of only one visit)
  The single stage treadmill test is a valid and easily performed submaximal test that estimates the VO2max of healthy adults aged 20-59 years. The test involves a 4 minute warm up at 0% grade at a self-selected walking speed that elicits a heart rate within 50-70% of the individual's age-predicted maximum heart rate.
6 Minute Walk Test | Single Study Visit (Study consists of only one visit)
  The test measures the distance that an individual can walk on a flat, hard surface in a period of 6 minutes. It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism.

SECONDARY OUTCOMES:
The Borg Rating of Perceived Exertion Scale (RPE) | Single Study Visit (Study consists of only one visit)
  The RPE scale measures feelings of effort, strain, discomfort and/or fatigue experienced during both aerobic and resistance training. It is based on the physical sensations a person experiences during physical activity, including increased heart rate, increased respiration or breathing rate, increased sweating, and muscle fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No